CLINICAL TRIAL: NCT04926389
Title: The Effect of Two Low-level Laser Irradiation Protocols on the Rate of Canine Retraction (a Randomized Controlled Clinical Trial)
Brief Title: Two Low-level Laser Irradiation Protocols on the Rate of Canine Retraction
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Hams Hamed Abdelrahman (Other)
Responsible Party: Sponsor-Investigator, Hams Hamed Abdelrahman, Assistant lecturer of DPH and Clinical statistician, Alexandria University
Organization: Alexandria University (Other)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: Canine retraction 2020
Record Dates: First submitted 2021-06-03; First posted 2021-06-15 (Actual); Last update posted 2021-06-15 (Actual); Status verified 2021-06

CONDITIONS: Malocclusion
MeSH Terms: conditions — Malocclusion

STUDY DESIGN:
Who Masked: Participant
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- low-level laser therapy applied on days 0, 3,7,14 & every 2 weeks (Experimental)
  Interventions: Other: low-level laser therapy applied on days 0, 3,7,14 & every 2 weeks
- low-level laser therapy applied every 3 weeks (Active Comparator)
  Interventions: Other: low-level laser therapy applied every 3 weeks

INTERVENTIONS:
Other: low-level laser therapy applied on days 0, 3,7,14 & every 2 weeks — one side of the maxillary arch will randomly receive LLLT on days 0, 3, 7, 14, and every 2 weeks thereafter and the contralateral side will serve as the controls.
  Arms: low-level laser therapy applied on days 0, 3,7,14 & every 2 weeks
Other: low-level laser therapy applied every 3 weeks — one side will also be randomly chosen to receive LLLT every 3 weeks and the contralateral side will serve as the controls.
  Arms: low-level laser therapy applied every 3 weeks

SUMMARY:
Several methods aiming at the acceleration of orthodontic tooth movement have been proposed, including low-level laser therapy (LLLT), which showed promising results. However, the frequency of patient recall has been one of its major drawbacks.

DETAILED DESCRIPTION:
A randomized controlled clinical trial will be conducted to address the aim of the study. Sixteen patients will be recruited, requiring the therapeutic extraction of the maxillary 1st premolars, with subsequent canine retraction into the extraction space. The sample will be randomly divided into 2 equal groups, each including 8 subjects.

In Group A, one side of the maxillary arch will randomly receive LLLT on days 0, 3, 7, 14, and every 2 weeks thereafter, while in Group B, one side will also be randomly chosen to receive LLLT every 3 weeks. The contralateral sides of both groups will serve as the controls. The LLLT applied will be Diode laser emitting infrared radiation at wavelength of 980 nm, in a continuous mode.

Canine retraction in both groups will be carried out bilaterally using nickel-titanium closed-coil spring, delivering 150 grams of force, and the rate of tooth movement will be checked every 3 weeks, over a period of 3 months. Other variables will be also examined including, interleukin-1β level in the gingival crevicular fluid, root resorption, and molar anchorage loss.

ELIGIBILITY:
Inclusion Criteria:

* Malocclusion requires at least the extraction of maxillary first premolars, followed by canine retraction into the extraction site.
* Normal shape and structure of the maxillary canines, with no history of root canal treatment.
* Patients with good oral hygiene, and a healthy periodontal condition.

Exclusion Criteria:

* Patients who underwent previous orthodontic treatment.
* Patients currently receiving drug therapy that may affect orthodontic tooth movement, e.g. hormonal therapy and corticosteroids.
* Patients with chronic diseases that may affect the rate of tooth movement.
* Pregnancy and lactation

Ages: 15 Years to 25 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 16 (Estimated)
Dates: Start 2020-01-01 (Actual); Primary Completion 2021-06-15 (Estimated); Study Completion 2021-06-15 (Estimated)

PRIMARY OUTCOMES:
Change in rate of canine retraction | at baseline and every 3 weeks for 3 months
  Several landmarks will be identified on the dental cast, including the mid-palatal raphe, the most medial points on the third right and left rugae, and the cusp tips of the right and left maxillary canines. Perpendicular lines will be drawn from the medial points of the right and left third rugae, and the cusp tips of the right and left maxillary canines to the mid-palatal raphe. The antero-posterior measurements will be carried out between the canine lines and the third rugae lines bilaterally, to assess the rate of canine retraction.
change in IL-1β level in the Ginigval Crevicular Fluid | at baseline, 7th, 17th and 21st day
  Samples from the GCF will be collected at baseline (before the first canine retraction), in addition to days 7, 14, and 21. GCF samples will be collected from the distal crevices of the canines, in Groups A and B, on both the experimental and control sides. Measurement of IL-1β level in the GCF will be performed using an ELISA kit.

SECONDARY OUTCOMES:
change canine root resorption: | at baseline and 3 months
  Root resorption of the maxillary canines will be evaluated and measured on the acquired pre-retraction and post-retraction CBCT scans.
Change molar anchorage loss | at baseline and every 3 weeks for 3 months
  Perpendicular lines will be drawn from the central fossae of both maxillary right and left first molars to the mid-palatal raphe. Consequently, molar anchorage loss will be calculated by measuring the distance between those lines, and the lines representing the third rugae as previously mentioned.

CONTACTS AND LOCATIONS:
Locations (1):
- Alexandria Faculty of Dentistry, Alexandria, Egypt

REFERENCES:
- [Derived] Eid FY, El-Kenany WA, Mowafy MI, El-Kalza AR. The influence of two photobiomodulation protocols on orthodontically induced inflammatory root resorption (a randomized controlled clinical trial). BMC Oral Health. 2022 Jun 5;22(1):221. doi: 10.1186/s12903-022-02251-w. PMID 35659655